CLINICAL TRIAL: NCT00123461
Title: A Phase 4, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Study to Assess the Efficacy and Safety of Doxercalciferol Capsules in Vitamin D-replete Subjects With Chronic Kidney Disease (CKD) Stages 3 or 4 With Secondary Hyperparathyroidism (SHPT).
Brief Title: Study of Safety and Efficacy of Doxercalciferol in Patients With Chronic Kidney Disease, Stage 3 or 4, and Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCI-CH-151
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Secondary Hyperparathyroidism; Renal Failure; Chronic Renal Insufficiency
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency; Renal Insufficiency, Chronic | interventions — 1 alpha-hydroxyergocalciferol

INTERVENTIONS:
Drug: Hectorol (doxercalciferol capsules), 0.5mcg

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of Hectorol® (doxercalciferol) capsules in treating patients with Stage 3 or Stage 4 chronic kidney disease (CKD) with secondary hyperparathyroidism who have vitamin D levels in the normal range. Previous studies with doxercalciferol were conducted in patients who had low levels of vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Plasma iPTH value above 110 pg/mL for CKD Stage 3 subjects or above 150 pg/mL for CKD Stage 4
* Serum 25-hydroxyvitamin D level greater than or equal to 30 ng/mL
* CKD Stage 3 evidenced by a glomerular filtration rate (GFR) from the abbreviated MDRD equation between 30-59 mL/min or CKD Stage 4 evidenced by a glomerular filtration rate (GFR) from the abbreviated MDRD equation between 15-29 mL/min

Exclusion Criteria:

* Serum cCa > 9.5 mg/dL
* Serum P > 4.6 mg/dL
* Abnormal liver functions
* Anticipated requirement for maintenance hemodialysis
* Use of active vitamin D sterol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Laboratory measurement of intact parathyroid hormone (iPTH) | 6 months

SECONDARY OUTCOMES:
Laboratory measurement of serum bone markers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (19):
- United States (17):
  - AKDHC Medical Research Services, Phoenix, Arizona
  - UCLA Diabetes Reseach Center, Alhambra, California
  - Apex Research of Riverside, Riverside, California
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Discovery Medical Research Group, Ocala, Florida
  - Nephrology Associates, Palm Beach Gardens, Florida
  - Georgia Kidney Associates, Inc., Marietta, Georgia
  - Michigan Kidney Consultants, P.C., Pontiac, Michigan
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Nephrology Associates, PA, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Altru Health System Research Center, Grand Forks, North Dakota
  - DaVita Lewiston Dialysis Center, Lewiston, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
- Puerto Rico (2):
  - Instituto Renal del Este, Caguas
  - Jose Cangiano, MD, San Juan

REFERENCES:
- See also: US FDA Approved Full Prescribing Information for Hectorol® Capsules — http://www.hectorol.com/docs/Hectorol%20Capsule%20PI%20Text_2006-01.pdf